CLINICAL TRIAL: NCT02204878
Title: A Randomized, Phase IV Study Exploring the Role of Parecoxib Sodium for Postoperative Pain Management in Open Hepatectomy
Brief Title: Role of Parecoxib Sodium for Postoperative Pain Management in Open Hepatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUMCH-Liver-Dynastat
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Hepatic Hemangioma Located in the Right Liver; Laparotomy Surgery
MeSH Terms: interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): 1ml of saline was given before anesthesia. PCA will be attached right before closing abdomen. Concentration of sufentanil is 1ug/ml. PCA settings: 1) no background infusion; 2) bolus 2ml sufentanil each; 3) with the lockout time 5 min, 1 hour limit: 10ml. 1ml saline Q12h will be given within 72 hours after surgery
- AT (Experimental): Dynastat 40mg was given before anesthesia. PCA will be attached right before closing abdomen. Concentration of sufentanil is 1ug/ml. PCA settings: 1) no background infusion; 2) bolus 2ml sufentanil each; 3) with the lockout time 5 min, 1 hour limit: 10ml. Dynastat 40mg Q12h will be given within 72 hours after surgery
  Interventions: Drug: Parecoxib Sodium

INTERVENTIONS:
Drug: Parecoxib Sodium — Dynastat 40mg was given before anesthesia. PCA will be attached right before closing abdomen. Concentration of sufentanil is 1ug/ml. PCA settings: 1) no background infusion; 2) bolus 2ml sufentanil each; 3) with the lockout time 5 min, 1 hour limit: 10ml. Dynastat 40mg Q12h will be given within 72 hours after surgery
  Arms: AT

SUMMARY:
To searching the role of parecoxib sodium for postoperative pain management in open hepatectomy

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-70 years old;
* Hepatic hemangioma patients who will undergo laparotomy surgery: diameter of hepatic hemangioma between 5-15cm, located in the right liver;
* Child score 5-6;
* BMI: 19-25;
* ASA: Ⅰ ~ Ⅱ grade;
* No comorbidities such as diabetes, hypertension, cardio renal or respiratory dysfunction, mental illness;
* No known allergies;
* No participation in other clinical trials within 2 months;
* Have been informed consent.
* Surgery-related: right subcostal incision, surgical time< 4 hours, hepatic pedicle occlusion time< 20 minutes, bleeding< 1000ml, no blood transfusions.

Exclusion Criteria:

* History of chronic pain，long-term use of analgesic drugs or alcohol abuse;
* Allergic to NSAIDs, opioids or sulfa drugs;
* Coagulopathy or other hematological disorder；
* Active peptic ulcer, gastrointestinal bleeding, inflammatory bowel disease;
* Pregnant or lactating;
* Mentally unstable to use PCA;
* Preoperative pain caused by other disease;
* Analgesic drugs or NSAIDs intake one week before surgery;
* Preoperative systemic inflammatory response syndrome;
* Preoperative chemotherapy or radiotherapy;
* Preoperative or postoperative use of steroids;
* Operative time> 4 hours, hepatic pedicle occlusion time> 20 minutes, blood loss> 1000ml, or intraoperative blood transfusion;
* TBil> 34 umol/L、PT prolongation> 3S、ALB< 30 g/L、or Child score> 7 within 42 hours after surgery；
* Bleeding、biliary fistula, intra-abdominal infections or other postoperative complications.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
VAS scores change | at rest and after activity befor and 6hrs, 18hrs, 30hrs, 42hrs, 54hrs and 66hrs after surgery

SECONDARY OUTCOMES:
liver function change | befor and 42hrs and 66hrs after surgery
kidney function change | befor and 42hrs and 66hrs after surgery
blood ammonia level change | before and 42hrs, 66hrs after surgery

OTHER OUTCOMES:
ESR change | before and 42hrs and 66hrs after surgery
portal blood flow change | before and after surgery
  Ultrasound evaluation
CRP change | before and 42hrs and 66hrs after surgery
IL4 change | before and 42hrs and 66hrs after surgery
IL6 change | before and 42hrs and 66hrs after surgery
portal blood pressure change | before and after surgery
  Ultrasound evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China